CLINICAL TRIAL: NCT07288788
Title: Assessment of Kidney Function in Patients With Epilepsy
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Hassan Ahmed, Resident Physician, Pediatrics, Sohag University
Other Study IDs: Soh-Med--25-9-2MS
Record Dates: First submitted 2025-11-21; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Observational study of pediatric patients admitted to Sohag University Hospital
  Interventions: Behavioral: Standard Clinical Observation

INTERVENTIONS:
Behavioral: Standard Clinical Observation — Observational study of pediatric patients admitted to Sohag University Hospital. No experimental treatment or device is administered. Data collection only.

SUMMARY:
This observational cross-sectional study aims to assess kidney function in pediatric patients with epilepsy attending Sohag University Hospital. The study evaluates renal biochemical markers, urinalysis, liver functions, abdominal ultrasonography, and the possible renal effects of long-term antiepileptic drug (AED) therapy.

DETAILED DESCRIPTION:
Epilepsy is one of the most common neurological disorders requiring long-term antiepileptic drug therapy. Many AEDs are metabolized hepatically but excreted renally, which may affect kidney function, especially with long-term use. Several AEDs-including topiramate, zonisamide, acetazolamide, carbamazepine, and valproate-have been associated with nephrolithiasis, tubular dysfunction, nephrotoxicity, and acute kidney injury.

The study evaluates renal function among children with idiopathic epilepsy using clinical assessment, laboratory markers (CBC, serum creatinine, electrolytes, ABG, urinalysis, liver functions), EEG findings, and abdominal ultrasound. The purpose is to estimate the prevalence of renal affection and its possible relation to AED use.

This observational cross-sectional study evaluates renal function in pediatric patients with epilepsy by measuring serum creatinine levels at the time of enrollment. The study will enroll children of various ages and both sexes, representing multiple epilepsy types and receiving different antiepileptic drug regimens.

Comprehensive baseline data, including demographic characteristics, medical history, seizure type and frequency, and current medication usage, will be collected. Venous blood samples will be obtained for serum creatinine measurement using validated clinical laboratory methods, ensuring standardized assessment of renal function.

The study's primary objective is to determine baseline renal function in this population and to investigate potential associations between antiepileptic drug therapy and renal outcomes. Secondary analyses will explore correlations between serum creatinine levels and patient-specific factors such as age, sex, epilepsy type, duration of therapy, and comorbidities.

All data will be handled in accordance with institutional and regulatory guidelines for clinical research. The results are intended to inform clinical monitoring practices, optimize antiepileptic drug management, and support future research on kidney function in children with epilepsy.

ELIGIBILITY:
Inclusion criteria

* Age: children between 1month and 15years old.
* Both sexes.
* children who suffering from idiopathic epilepsy

Exclusion criteria:

* Age: children below 1month old& children above 15 years old.
* Children suffer from convulsions due to CNS infection
* Children with non idiobathic epilepsy

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients admitted to Sohag University Hospital. Observational data will be collected from medical records.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-28 (Actual); Primary Completion 2025-09-28 (Actual); Study Completion 2026-09-28 (Estimated)

PRIMARY OUTCOMES:
Serum creatinine level in pediatric epilepsy patients | At enrollment (single cross-sectional assessment)
  Measurement of serum creatinine in pediatric patients at enrollment to assess renal function related to epilepsy or antiepileptic drug use

SECONDARY OUTCOMES:
Prevalence of nephrolithiasis / nephrocalcinosis | At enrollment (single cross-sectional assessment)
  Presence of renal calculi or nephrocalcinosis detected by abdominal ultrasound performed at enrollment.
Electrolyte disturbances | At enrollment (single cross-sectional assessment)
  Frequency of clinically significant electrolyte abnormalities (e.g., hypokalemia, hypernatremia, bicarbonate reduction) measured in serum chemistry at enrollment.
Abnormal urinalysis findings | At enrollment (single cross-sectional assessment)
  Proportion of participants with abnormal urine analysis results (proteinuria, hematuria, crystalluria, or other abnormalities) at enrollment.
Association between AED regimen and renal parameters | At enrollment (single cross-sectional assessment)
  Comparison of renal function markers (serum creatinine, urinalysis, ultrasound findings) across groups defined by type of antiepileptic drug(s) used (e.g., renally excreted vs. non-renally excreted drugs) at enrollment.
Abdominal Ultrasound Findings | At enrollment (single cross-sectional assessment)
  Detection of renal structural abnormalities including nephrolithiasis or nephrocalcinosis.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Sohag University, Sohag
  - Sohage Faculty of Medicine, Sohag

IPD SHARING:
Plan to Share IPD: Yes